CLINICAL TRIAL: NCT07094464
Title: A Single-Arm, Open-Label Phase I Clinical Study of Selinexor Combined With Azacitidine for Maintenance Therapy in TP53 Mutant AML/MDS Patients Post-Transplant
Brief Title: Maintenance Therapy With Selinexor and Azacitidine in TP53 Mutant AML/MDS After Transplantation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daihong Liu (Other)
Responsible Party: Sponsor-Investigator, Daihong Liu, Dr., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2025-055-01
Record Dates: First submitted 2025-06-01; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: TP53-mutated MDS and AML; Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: TP53 mutant myeloid tumors; allogeneic hematopoietic cell transplantation.
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Maintenance; selinexor; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assigned Interventions (Experimental): 1）Treatment will begin approximately 3 months post-transplant. The study duration will be 1 year with treatment cycles every 3 months, totaling 4 cycles.
  1. Selinexor: Single-arm phase I study with sequential dose escalation of Selinexor.
     Three dose levels will be tested in separate cohorts:
     * Cohort 1: Selinexor, 20 mg, twice a week for 2 weeks
     * Cohort 2: Selinexor, 40 mg, twice a week for 2 weeks
     * Cohort 3: Selinexor, 60 mg, twice a week for 2 weeks
  2. Azacitidine: 35 mg/m² for 5 days. 2）Bone marrow morphology, characteristic gene mutation or fusion gene quantification, immunophenotyping, chimerism, or transplant-related FISH will be assessed before and after each treatment cycle, according to the follow-up schedule post-transplant. Patients with hematological relapse at any time will discontinue from the experimental group and receive an alternative treatment.
  Interventions: Drug: Maintenance Therapy with Selinexor and Azacitidine

INTERVENTIONS:
Drug: Maintenance Therapy with Selinexor and Azacitidine — 1. Selinexor: Oral administration in 4 cycles:
     - Dose Escalation Phase: Cohort 1: Selinexor, 20 mg, twice a week for 2 weeks Cohort 2: Selinexor, 40 mg, twice a week for 2 weeks Cohort 3: Selinexor, 60 mg, twice a week for 2 weeks
     - Dose Expansion: MTD/RP2D will be determined based on safety.
  2. Azacitidine: 35 mg/m² for 5 days.

SUMMARY:
This study aims to explore the safety and efficacy of selinexor combined with azacitidine for maintenance therapy in TP53 mutant AML/MDS patients following transplantation.

DETAILED DESCRIPTION:
This research targets high-risk recurrence patients with TP53 mutations in AML/MDS, administering low-dose azacitidine combined with selinexor for maintenance treatment post-allo-HCT (Allogeneic Hematopoietic Cell Transplantation). The goal is to observe the safety and tolerability of this drug combination as maintenance therapy post-transplant. The primary outcome measure will be post-transplant recurrence rate and non-relapse survival rate, while secondary outcomes include overall survival and non-relapse mortality. Previous studies have indicated that azacitidine and selinexor are safe and effective in maintenance therapy for AML/MDS. This study aims to reduce the risk of recurrence and prolong disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* (1) Voluntary participation in the clinical study: Participant or legal guardian understands and signs the Informed Consent Form (ICF) and is willing to comply with all trial procedures.

  (2) Age below 75 years at screening; gender not restricted. (3) Diagnosed with AML or MDS with TP53 mutation (VAF ≥ 2%) and post-allo-HCT. (4) No severe allergic constitution. (5) Liver function: ALT and AST ≤ 2.5 times the upper limit of normal, bilirubin ≤ 2 times the upper limit of normal.

  (6) Renal function: creatinine ≤ upper limit of normal. (7) No uncontrolled infections or severe psychiatric disorders. (8) ECOG performance score of 0-3; life expectancy of 4 months or more. (9) Peripheral blood counts for granulocytes and platelets.

Exclusion Criteria:

* (1) Patients with known allergies or contraindications to the study drugs. (2) Pregnant or breastfeeding women. (3) Patients with uncontrolled active infections or active GVHD. (4) Patients with a long history of smoking or alcohol abuse affecting trial outcome evaluation.

  (5) Patients with psychiatric disorders or conditions preventing informed consent, unable to comply with treatment and assessment requirements.

  (6) Patients who underwent major surgery on important organs less than 6 weeks prior.

  (7) Abnormal liver function: ALT or AST > 2.5 times the upper limit of normal; bilirubin > 2 times the upper limit of normal; renal function: creatinine > upper limit of normal.

  (8) Patients deemed unsuitable for this clinical trial by the investigator (e.g., poor compliance, substance abuse).

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease relapse | 1 year after transplantation
  The definition of disease relapse: After remission, patients present with one of the following three conditions: (1) ≥5% of primary lymphocytes and immature lymphocytes in the bone marrow; (2) Extramedullary leukemia occurs; (3) Leukemia cells were found in peripheral blood smears. The definition of MRD recurrence: Leukemia cells are detected by flow cytometry or molecular biology.

SECONDARY OUTCOMES:
Non-relapse mortality (NRM) | 1 year after transplantation
  From the first day after stem cell infusion to the last follow-up time, the number of NRM patients/the total number of cases ×100%. Death not caused by recurrence in the CR state.
Overall survival (OS) | 1 year after transplantation
  The time from transplantation to death of any cause or the last follow-up day.
Progress-free survival (PFS) | 1 year after transplantation
  The time from the date of transplantation to the recurrence of leukemia or death for any reason.
Drug-related adverse events | 1 month after the last maintenance treatment ends
  All adverse events with a causal relationship to the study intervention (Selinexor + Azacitidine), assessed by investigators according to CTCAE v5.0 criteria.
Measurable Residual Disease (MRD) in bone marrow | 1 year after transplantation
  Quantitative assessment of residual leukemic cells using: FCM-MRD and TP53 mutation NGS testing

CONTACTS AND LOCATIONS:
Overall Officials: Dai-hong Liu, Dr., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data contain sensitive personal health information

REFERENCES:
- [Background] Mishra A, Tamari R, DeZern AE, Byrne MT, Gooptu M, Chen YB, Deeg HJ, Sallman D, Gallacher P, Wennborg A, Hickman DK, Attar EC, Fernandez HF. Eprenetapopt Plus Azacitidine After Allogeneic Hematopoietic Stem-Cell Transplantation for TP53-Mutant Acute Myeloid Leukemia and Myelodysplastic Syndromes. J Clin Oncol. 2022 Dec 1;40(34):3985-3993. doi: 10.1200/JCO.22.00181. Epub 2022 Jul 11. PMID 35816664
- [Background] Sakabe K, Nishikado A, Wakatsuki T, Oki T, Ito S. Right atrial potential profiles during atrial fibrillation predict the success of atrial defibrillation. J Electrocardiol. 1998 Jan;31(1):39-44. doi: 10.1016/s0022-0736(98)90005-x. PMID 9533376
- [Background] Santini V, Stahl M, Sallman DA. TP53 Mutations in Acute Leukemias and Myelodysplastic Syndromes: Insights and Treatment Updates. Am Soc Clin Oncol Educ Book. 2024 Jun;44(3):e432650. doi: 10.1200/EDBK_432650. PMID 38768424
- [Background] Peng F, Chen Nan-xian. Amplification of the interface-phonon population under an intense laser field. Phys Rev B Condens Matter. 1992 Sep 15;46(12):7627-7631. doi: 10.1103/physrevb.46.7627. No abstract available. PMID 10002503
- [Background] Najima Y. Overcoming relapse: prophylactic or pre-emptive use of azacitidine or FLT3 inhibitors after allogeneic transplantation for AML or MDS. Int J Hematol. 2023 Aug;118(2):169-182. doi: 10.1007/s12185-023-03596-w. Epub 2023 Apr 10. PMID 37036626
- [Background] Lutz S. Columbia/HCA backs hospital's expansion. Mod Healthc. 1994 Aug 29;24(35):42. No abstract available. PMID 10136154
- [Background] Berkhout TA, Gohil J, Gonzalez P, Nicols CL, Moores KE, Macphee CH, White JR, Groot PH. Selective binding of the truncated form of the chemokine CKbeta8 (25-99) to CC chemokine receptor 1(CCR1). Biochem Pharmacol. 2000 Mar 1;59(5):591-6. doi: 10.1016/s0006-2952(99)00354-8. PMID 10660125
- [Background] Minowa M, Orito S, Tsuchiaki M, Tsukamoto T. Search for resonances in the e+e---> gamma gamma process in the mass region around 1.062 MeV/c2. Phys Rev Lett. 1989 Mar 6;62(10):1091-1094. doi: 10.1103/PhysRevLett.62.1091. No abstract available. PMID 10039574
- [Background] Reading NS, Aust SD. Engineering a disulfide bond in recombinant manganese peroxidase results in increased thermostability. Biotechnol Prog. 2000 May-Jun;16(3):326-33. doi: 10.1021/bp0000151. PMID 10835231
- [Background] Masuda Y, Sadato D, Toya T, Hosoda Y, Hirama C, Shimizu H, Najima Y, Harada H, Harada Y, Doki N. Transplantation outcomes of TP53-mutant AML and MDS: a single transplantation center experience of 63 patients. Int J Hematol. 2025 Jun;121(6):820-832. doi: 10.1007/s12185-025-03951-z. Epub 2025 Feb 26. PMID 40011351